CLINICAL TRIAL: NCT06378528
Title: A Preliminary Trial of Safety and Feasibility of Ketamine-assisted Psychotherapy in Adolescents With Posttraumatic Stress-disorder
Brief Title: Ketamine-assisted Psychotherapy for Adolescent PTSD (KAP)
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Budgeting/funding
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1706; Protocol Version 11/14/25 (Other: UW Madison); A538900 (Other: UW Madison)
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-08

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: single group, open label, pilot study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adolescents with Severe PTSD (Experimental)
  Interventions: Drug: Ketamine; Device: SmartSleep EEG recording headband

INTERVENTIONS:
Drug: Ketamine — 3 Intravenous ketamine administrations (0.5mg/kg, not to exceed 40mg dose) immediately prior to a psychotherapy session over the span of 6 weeks
  Other Names: Ketamine Assisted Psychotherapy
Device: SmartSleep EEG recording headband — Participants will complete 7 nights of at-home sleep recordings for exploratory analysis

SUMMARY:
The objectives of this study are to investigate the feasibility, tolerability, and preliminary efficacy of repeated ketamine-assisted psychotherapy sessions in adolescents with severe posttraumatic stress disorder. The study will enroll adolescents with a current diagnosis of posttraumatic stress disorder (PTSD) to complete three intravenous ketamine administrations accompanied by a psychotherapy session over the span of six weeks. All participants will complete an initial set of preparatory sessions, and each dosing session will be followed by three to six hours of integration sessions. Finally, participants will complete 7 nights of at-home sleep recordings. The investigators hypothesize that this protocol will be well-tolerated by adolescents and that patients will experience decreases in PTSD symptom severity at follow-up.

DETAILED DESCRIPTION:
Primary Objective:

* Characterize safety and adverse events associated with repeated ketamine-assisted psychotherapy in adolescents with PTSD.

Secondary Objectives:

* Evaluate initial feasibility of recruitment and retention of adolescents with PTSD.
* Explore potential impacts of ketamine-assisted psychotherapy on PTSD symptom severity at follow-up

ELIGIBILITY:
Inclusion Criteria:

* Aged 15-17 years old, inclusive
* At baseline, meet threshold for Diagnostic and Statistical Manual (DSM-5) criteria for current PTSD as determined by the CAPS-CA.
* Medically and neurologically healthy on the basis of physical examination, medical history, and the clinical judgement of the evaluating study medical provider
* Must agree to inform the investigators within 48 hours of any emergent medical conditions and procedures
* If of childbearing potential, must have a negative pregnancy test at study entry and prior to each KAP dosing session, and must agree to use adequate birth control through 10 days after the last KAP dosing session.
* Must agree not to participate in any other interventional clinical trials during the duration of the study
* Must be willing to comply with all study procedures
* A primary parent or guardian is willing to provide informed consent
* Are fluent in or predominantly speaking and reading in English

Exclusion Criteria:

* Caregiver or adolescent is unwilling or unable to give adequate informed consent
* Are likely, in the investigator's opinion and via observation during the Preparatory Period, to be re-exposed to their index trauma or other significant trauma, lack social support, or lack a stable living situation during study participation.
* Any finding(s), based on the screening process, that the PI feels would make the study unsuitable for the participant.
* Current diagnosis of or history of a psychotic disorder, bipolar disorder, or autism spectrum disorder diagnosed by the Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS) interview and clinician judgement. No other co-morbid disorders are exclusionary.
* Intellectual disability (IQ<70) per medical history
* History of moderate to severe substance use disorder, as determined by the KSADS and/or clinician judgement (excluding tobacco), or active substance use (including current alcohol use or positive urine toxicology)
* Any prior exposure to sub-anesthetic doses of ketamine (including prior research or clinical psychiatric treatment with ketamine and/or recreational use)
* Any participant presenting current serious suicide risk, as determined through the KSADS, responses to Columbia Suicide Severity Rating Scale (C-SSRS), and/or clinical judgment of the investigator, will be excluded; however, history of suicide attempts prior to enrollment is not an exclusion.
* Would present a serious risk to others as established through clinical interview and contact with treating physician.
* Current use benzodiazepines, opiates, or lamotrigine, which are hypothesized to interfere with ketamine's mechanism of action
* High blood pressure (BP) at the time of screening, defined by the Centers for Disease Control and Prevention (CDC) to be BP greater than 130/80.
* Persons who have previously received ketamine therapeutically or taken it recreationally.
* Are pregnant, nursing, or are able to become pregnant and are not practicing an effective means of birth control.
* Persons who are known to have a hypersensitivity to ketamine
* Participants that are deemed not to be medically and neurologically healthy on the basis of physical examination, medical history, and the clinical judgement of the Study Medical Provider or qualified designee in order to participate.

  * Examples of medical rule-outs include but are not limited to: unstable hypertension, recent severe neurologic injury, a history or current signs/symptoms of liver or renal insufficiency, and current diagnoses of cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disorders that are deemed clinically significant based on investigator judgement.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Summary of Adverse Events Attributable to Ketamine Administration | through the last study visit, up to 10 weeks
  Degree of adverse effects (AEs) attributable to ketamine administration as categorized according to the abbreviated (six-item) Clinician-Administered Dissociative States Scale (CADSS-6), which assesses situation-dependent dissociative states, and the Systematic Assessment for Treatment Emergent Events (SAFTEE-GI), which uses a standardized general (SAFTEE-GI) inquiry of physical/health problems and possible treatment-emergent side effects. The SAFTEE-GI will be administered during the preparatory period, at every KAP dosing session, integration, and endpoint assessment visit, the CADSS-6 will be administered at every KAP dosing session and during each integration period. Reported here are a list of AEs attributed to KAP Administration with count of participants experiencing them.

SECONDARY OUTCOMES:
Number of Participants Adhering to the Study Protocol | up to 10 weeks
  Study protocol adherence for preparation, dosing, and follow-up visits.
Number of Visits Completed Throughout the Study Duration | up to 10 weeks
  There are approximately 16 study visits from screening through one month follow up.

OTHER OUTCOMES:
Changes in PTSD symptom severity as measured by the Clinician Administered PTSD Scale Child/Adolescent Version (CAPS-CA) | baseline and 1 month follow up (at up to 10 weeks on study)
  The CAPS-CA is a well-validated instrument in adolescent populations and is used often in pediatric clinical trials. This outcome will assess the current severity of overall PTSD symptomatology. Assessments of this endpoint will occur prior to any preparatory sessions and again at a 1-month follow-up. Scores indicate a PTSD severity rating from 0 (absent), 1 (mild), 2 (moderate), 3 (severe), or 4 (extreme).
Exploratory Measurements: Change waveform recorded with Philips SmartSleep headband, measured in Hz | 7 consecutive nights surrounding the first KAP session, during study week 2
  During the first KAP session week, sleep will be recorded for seven nights (3 nights prior to the KAP session, night of KAP session, and 3 nights after KAP session) using the Philips SmartSleep recording headband. The SmartSleep device collects real-time EEG data. The EEG signals are acquired at 1000 Hz, high-pass filtered using a single pole filter (0.3 Hz cutoff frequency), notch filtered at 50 Hz and 60 Hz to remove power-line noise, and down-sampled to 250 Hz for real-time, onboard sleep scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nicholas, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No